CLINICAL TRIAL: NCT05060536
Title: Infrapatellar Fat Pad Excision in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 299830
Record Dates: First submitted 2021-09-15; First posted 2021-09-29 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Knee Discomfort; Arthroplasty Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removal of infrapatellar fat pad (Active Comparator): When patients will have their fat pad removed.
  Interventions: Procedure: Removal of infrapatellar fat pad
- No removal of infrapatellar fat pad (Placebo Comparator): When patients will not have their fat pad removed.
  Interventions: Procedure: No removal of infrapatellar fat pad

INTERVENTIONS:
Procedure: Removal of infrapatellar fat pad — There is no agreed protocol for retaining or excising the infrapatellar fat pad with many surgeons routinely completely removing the fat pad to improve view of the proximal tibia while others opt to retain or minimally excise the tissue.
  We are aware of no risks involved in performing this procedure and current practice of many orthopaedic surgeons is either to routinely remove or routinely retain the infrapatellar fat pad when performing total knee arthroplasty.
  The potential benefits are that we will understand better whether removing or retaining this tissue does have a role in influencing outcomes after total knee replacement surgery. The results will be disseminated to the wider orthopaedic community to inform practice with the aim or improving outcomes from total knee arthroplasty.
  Arms: Removal of infrapatellar fat pad
Procedure: No removal of infrapatellar fat pad — Retaining the infrapatellar fat pad during total knee replacement- no surgical removal.
  Arms: No removal of infrapatellar fat pad

SUMMARY:
To examine whether removing the infrapatellar fat pad from the knee during total knee arthroplasty affects the patient outcome in terms of pain and knee function following the procedure. Currently there is no consensus on whether removing this tissue from the knee has a positive or detrimental effect. Small studies have been published, some showing improved symptoms and some worse symptoms. Current practice of orthopaedic surgeons is either to routinely remove or routinely retain the tissue when performing total knee arthroplasty.

DETAILED DESCRIPTION:
Aim and Objectives The aim of the study is to examine whether removing or retaining the infrapatellar fat pad influences pain or knee function in the short and medium term.

Study Design A single centre randomized controlled trial of total knee arthroplasty with and without infrapatellar fat pad excision

Methodology A research nurse or the responsible consultant orthopaedic surgeon will identify potentially eligible patients from the list of those invited to attend the pre-operative assessment clinic for total knee arthroplasty. As part of their written invitation to attend this clinic, they will receive an information leaflet about the study from their consultant.

A research nurse or the responsible consultant orthopaedic surgeon will discuss the trial with them at the pre-assessment clinic. If the patient is willing to take part in the study they would then be asked to sign a consent form and will be reminded of the opportunity to withdraw from the study at any point. Their consent will be confirmed on the day of their admission for surgery.

Consented patients will be randomized to one of two arms of the study, the only variable being whether or not the infrapatellar fat pad is excised.

Randomisation to excision or retention of the infrapatellar fat pad will occur immediately prior to the total knee arthroplasty procedure being performed, and will be performed using the program freely available at http://www.randomization.com. Sealed envelopes will be prepared and the operating surgeon will open the randomisation envelope immediately before performing the total knee arthroplasty procedure. The procedure will then be performed and recorded. The excision of the infrapatellar fat pad itself takes less than 20 seconds to perform, and the knee replacement procedure is otherwise performed as normal. The outcome of the randomisation and procedure performed will be known only to the operating surgeon and researcher and not to those following up the patients and recording the outcome measures.

Seven consultant orthopaedic surgeons will take part in the trial. All perform total knee arthroplasty surgery regularly . Other than the consent process and additional questionnaires and clinical assessment performed, the care of patients in the study will be identical to all other non-study patients. Follow up will follow our normal routine pathway of visits at 3 months, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male/female patients between 40 and 100 years of age
* Undergoing primary total knee arthroplasty

Exclusion Criteria:

* Patient undergoing unicompartmental knee arthroplasty
* Patient undergoing revision knee arthroplasty
* Patient undergoing arthroplasty using non standard implants
* Previous patella surgery or injury
* Cognitive impairment
* Lack of conversational English

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Knee pain | 3 months post-operatively
  As assessed by patient reported outcome scores: Oxford knee score (0-48) Higher score better outcome.
Knee pain | 1 year post-operatively
  As assessed by patient reported outcome scores: Oxford knee score (0-48) Higher score better outcome.
Knee pain | 2 years post-operatively
  As assessed by patient reported outcome scores: Oxford knee score (0-48) Higher score better outcome.
Knee pain (Anterior) | 3 months post-operatively
  As assessed by patient reported outcome scores: Kujala score (0-100) Higher score better outcome.
Knee pain (Anterior) | 1 year post-operatively
  As assessed by patient reported outcome scores: Kujala score (0-100) Higher score better outcome.
Knee pain (Anterior) | 2 years post-operatively
  As assessed by patient reported outcome scores: Kujala score (0-100) Higher score better outcome.
Knee function | 3 months post-operatively
  As assessed by patient reported outcome scores: Oxford knee score (0-48) Higher score better outcome.
Knee function | 1 year post-operatively
  As assessed by patient reported outcome scores: Oxford knee score (0-48) Higher score better outcome.
Knee function | 2 years post-operatively
  As assessed by patient reported outcome scores: Oxford knee score (0-48) Higher score better outcome.

SECONDARY OUTCOMES:
Knee Range of Movement- flexion and extension in degrees | 3 months post-operatively
  Measured in degrees with goniometer
Knee Range of Movement- flexion and extension in degrees | 1 year post-operatively
  Measured in degrees with goniometer
Knee Range of Movement- flexion and extension in degrees | 2 years post-operatively
  Measured in degrees with goniometer
Shortening of patellar tendon- comparison between X-ray at 3 months with pre-operative X-ray | 3 months post-operatively
  Measured on X-ray in millimeters
Shortening of patellar tendon- comparison between X-ray at 1 year with pre-operative X-ray | 1 year post-operatively
  Measured on X-ray in millimeters
Shortening of patellar tendon- comparison between X-ray at 2 years with pre-operative X-ray | 2 years post-operatively
  Measured on X-ray in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Simon Spencer, MBBS. FRCS., Study Director — NHS Greater Glasgow and Clyde Board HQ
Locations (1):
- NHS Greater Glasgow and Clyde. Queen Elizabeth hospital (Victoria & Gartnavel), Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No